CLINICAL TRIAL: NCT02336061
Title: Evaluation of Gender Differences on the Psychosocial and Economic Impact in Patients With Advanced Non-small Cell Lung Cancer.
Acronym: IMPULSO
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision due to the low recruitment rate
Sponsor: Asociación para la Investigación del Cáncer de Pulmón en Mujeres (Other)
Collaborators: Pivotal S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: ICA-QUI-2014-01
Record Dates: First submitted 2014-12-03; First posted 2015-01-12 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- male: It will be stratified based on biological sex, age and smoking to guarantee homogeneity between the cohorts.
  Interventions: Behavioral: Evaluation of gender differences on the psychosocial and economic impact.
- female: It will be stratified based on biological sex, age and smoking to guarantee homogeneity between the cohorts.

INTERVENTIONS:
Behavioral: Evaluation of gender differences on the psychosocial and economic impact.
  Groups: male

SUMMARY:
The purpose of this study is to evaluate of gender differences on the psychosocial and economic impact in patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
Multi-centre, prospective follow-up post-authorisation study of two patient cohorts with metastatic NSCLC (men and women). It will be stratified based on biological sex, age and smoking to guarantee homogeneity between the cohorts. The clinical procedures for assessing the tumour and the treatment response will be performed according to the site's standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage IV NSCLC who are going to commence first line treatment
* Patients over the age of 18
* ECOG 0-3
* Patients who have granted their informed consent, preferably in writing, but otherwise, verbal with witnesses who are independent of the research team
* Life expectancy of over three months
* Speak fluent Spanish, in order to be able to complete the study questionnaires
* Patients able to read and write with no problems

Exclusion Criteria:

* Previous systemic treatment for metastatic NSCLC. The administration of neoadjuvant or adjuvant radiotherapy and/or chemotherapy is permitted provided it was completed major or equal 6 months prior
* Dementia or a significantly altered mental state that could affect comprehension or the ability to grant informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1250 patients over 18 years of age (approximately 50% men/women), with metastatic NSCLC, who are going to commence first-line treatment and who have a life expectancy of over three months will be included. They will be distributed into two cohorts (men and women) at 50% and will be distributed by age group and smoking status to facilitate the homogeneity between the two cohorts.
Sampling Method: Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Psychosocial impact (Test Family APGAR, Partner Test and adapted Duke-UNC-11 Scale) | 2 years
  The procedures for assessing psychosocial impact are: Test Family APGAR, Partner Test and adapted Duke-UNC-11 Scale. These tests will be performed by the investigator at visit baseline, visit 2 visit 3 and visit 4, according to the site's standard practice until patient death or for up to 24 months from the time of inclusion.
Economic impact (employment status, working hours, income range, public assistance, family support ...) | 2 years
  The procedures for assessing economic impact are some specific economic variables (employment status, working hours, income range, public assistance, family support ...)

SECONDARY OUTCOMES:
Influence of treatment (reatment received, treatment received, tumour ssessment, Medical history, including history of smoking, ECOG performance status, associated medical conditions and prior treatments administered (surgery, adjuvant treatment). | 2 years
  The procedures for assessing to influence of treatment are:Treatment received, treatment received, tumour ssessment, Medical history, including history of smoking, ECOG performance status, associated medical conditions and prior treatments administered (surgery, adjuvant treatment). These will be performed in line with the site's standard practice at visit baseline, visit 2 visit 3 and visit 4, according to the site's standard practice until patient death or for up to 24 months from the time of inclusion.
Psychosocial and economic impact on the primary caregiver (Zarit Caregiver Burden Questionnaire and Test assessing the economic impact) | 2 years
  The procedures for assessing psychosocial and economic impact are: Zarit Caregiver Burden Questionnaire and Test assessing the economic impact. These will be performed in line with the site's standard practice at visit baseline, visit 2 visit 3 and visit 4, according to the site's standard practice until patient death or for up to 24 months from the time of inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: María Rosario García, MD, Study Chair — Complejo Hospitalario A Coruña; Pilar Garrido, MD, Study Chair — Hospital Universitario Ramón y Cajal; Nuria Viñolas, MD, Study Chair — Hospital Clinic of Barcelona
Locations (18):
- Spain (18):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital de Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital German Trias i Pujol, Badalona, Barcelona
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Arnau de Villanova, Valencia
  - Hospital La Fe, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Vinolas NN, Garcia-Campelo R, Majem M, Carcereny E, Isla D, Gonzalez-Larriba JL, Coves J, De-Castro J, Domine M, Lianes P, Artal A, Remon J, Felip E, Garrido P. Assessment of the psychosocial and economic impact according to sex in non-small cell lung cancer patients: an exploratory longitudinal study. BMC Psychol. 2020 Nov 23;8(1):123. doi: 10.1186/s40359-020-00489-z. PMID 33228796